CLINICAL TRIAL: NCT00395941
Title: Efficacy and Safety of Acitretin Plus Pioglitazone in Patients With Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, SHotra, professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pharma 6/699
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Pioglitazone; Acitretin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Acitretin
  Interventions: Drug: Acitretin
- Experimental (Experimental): Pioglitazone
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone
  Arms: Experimental
Drug: Acitretin — Acitretin
  Arms: Control

SUMMARY:
Acitretin, when given in combiantion with pioglitazone might achieve better and/or more rapid control of moderate to severe chronic plaque type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic plaque type psoriasis having body surface area involvement of > 20%
* Patients of either sex
* Females who have completed their family and are tubectomized or are postmenopausal i.e. no menstrual bleeding over at least 1 year
* Age range 18-65 years

Exclusion Criteria:

* Females of child bearing potential
* H/O hypersensitivity to acitretin
* Impaired hepatic function (serum bilirubin, AST, ALT and alkaline phosphatase >1.5 times the upper limit of normal)
* Impaired renal function (serum creatinine >1.5mg% in males and >1.4 mg% in females)
* Hyperlipidemia
* BMI >30 kg /m2
* H/O excessive alcohol use
* Diabetes mellitus
* Congestive heart failure
* Ischemic heart disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in PASI score from baseline in the two groups | 12 weeks

SECONDARY OUTCOMES:
Proportion of subjects with an improvement of at least 75% in the psoriasis area-and-severity index (PASI) by week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Dogra, MD, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, India

REFERENCES:
- [Derived] Mittal R, Malhotra S, Pandhi P, Kaur I, Dogra S. Efficacy and safety of combination Acitretin and Pioglitazone therapy in patients with moderate to severe chronic plaque-type psoriasis: a randomized, double-blind, placebo-controlled clinical trial. Arch Dermatol. 2009 Apr;145(4):387-93. doi: 10.1001/archdermatol.2009.5. PMID 19380660